CLINICAL TRIAL: NCT01377649
Title: Contrast Ultrasound Perfusion Imaging in Peripheral Arterial Disease
Brief Title: Contrast Ultrasound Perfusion Imaging in Peripheral Arterial Disease (PAD)
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: IRB00007524
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Age matched control subjects without PAD
- Patients with PAD

SUMMARY:
Contrast ultrasound is a technique that can quantify blood flow in the tissues of the body by ultrasound detection of microbubble contrast agents that behave in the circulation similar to red blood cells. In this study, the investigators hypothesize that contrast ultrasound of blood flow in the leg (thigh and calf) at rest and during stress produced by medications that mimic exercise (vasodilator stress) can provide information on the location and severity of peripheral vascular disease (blockages of the blood vessels in the leg). The investigators will also determine whether symptom improvement after revascularization (procedures to open up or bypass the blockages) is directly related to the improvement in blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Known or suspected PAD
2. Lower extremity angiography or MRA planned or performed within 6 months

Exclusion Criteria:

1. Age <19 y.o.
2. Pregnant or lactating females
3. Hypersensitivity to ultrasound contrast agent, dipyridamole, or regadenoson
4. Severe reactive airways disease
5. Evidence right-to-left shunt (identified on screening echo)
6. NYHA Class III or IV heart failure.
7. Planned amputation
8. Unstable coronary artery disease or severe aortic stenosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease who are referred for diagnostic angiography and/or revascularization procedures
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Quantitation of Perfusion | Immediate
  Correlation of skeletal muscle perfusion with symptom status

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States